CLINICAL TRIAL: NCT04408404
Title: Factors Influencing Perioperative Mortality in Type A Acute Aortic Dissections Operated at Dijon University Hospital
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier La Chartreuse (Other)
Responsible Party: Principal Investigator, MORGANT Marie-Catherine, Principal investigator, Centre Hospitalier La Chartreuse
Other Study IDs: CCVT- Dissection
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type A aortic dissection: Patient operated for type A acute aortic dissection between 01 January 2007 and 31 December 2017 in Dijon Burgundy University Hospital
  Interventions: Procedure: Acute aortic dissection

INTERVENTIONS:
Procedure: Acute aortic dissection — Acute aortic dissection treatment include Bentall procedure, Tyrone David procedure, Yacoub procedure or ascendant aortic replacement with or without aortic valve replacement, ascendant aortic root remodelling (all are standard of care procedures)

SUMMARY:
Type A acute aortic dissections are a rare condition whose natural evolution is catastrophic. Global mortality remains high even if it decreased last years. This is probably due to improvement of diagnostic techniques and the evolution of surgical practices. It is however important to have medical data and statistics obtained in past years in order to better understand the factors influencing peroperative mortality and thereby to continue this improvement.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent aortic dissection surgery in Dijon Burgundy University Hospital

Exclusion Criteria:

* patients who died before the surgical incision

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent aortic dissection surgery in Dijon Burgundy University Hospital since the 01 January 2007 and the 31 december 2017.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Monitor peri-operative mortality incidence rates | 1 day
  Mortality during peri-operative acute aortic dissection procedure

SECONDARY OUTCOMES:
Monitor peri-operative morbidity incidence rates | 1 day
  Stroke, Kidney failure, Reexploration for bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular and thoracic surgery Unit - Dijon University Hopital, Dijon, France

IPD SHARING:
Plan to Share IPD: No
All patients are informed before surgery that all the medical data included in the medical record could be used in cardiovascular monocentric retrospective study. No data shared.